CLINICAL TRIAL: NCT06825585
Title: Efficacy and Visual Quality of Orthokeratology Lenses With Different Designs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xiaoyan Yang (Other)
Responsible Party: Sponsor-Investigator, Xiaoyan Yang, Tianjin Eye Hospital, Tianjin Eye Hospital
Organization: Tianjin Eye Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Different Orthk lens
Record Dates: First submitted 2025-02-09; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Myopia; Myopia; Refractive Error
MeSH Terms: conditions — Myopia; Refractive Errors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Myopic children who need OK lens treatment
  Interventions: Device: Orthokeratology with 5.0mm back optical zone diameter
- Control group (Active Comparator): Myopic children who need OK lens treatment
  Interventions: Device: Orthokeratology with a 6.2 mm back optical zone diameter

INTERVENTIONS:
Device: Orthokeratology with 5.0mm back optical zone diameter — The orthokeratology lenses used in this study were Double Reservoir Lenses (DRL) manufactured by Precilens (Creteil, France). The lenses feature a dual reverse-curve design with a back optic zone diameter (BOZD) of 5.0 mm.
  Arms: Experimental Group
Device: Orthokeratology with a 6.2 mm back optical zone diameter — The orthokeratology lenses used were Euclid lenses manufactured by Euclid Systems (Herndon, VA, USA). These lenses feature a four-zone, five-curve design with a back optic zone diameter (BOZD) of 6.2 mm.
  Arms: Control group

SUMMARY:
Orthokeratology (ortho-k) lens is very effective in slowing down axial elongation in myopic children by 30% to 63% when compared to children wearing single-vision spectacles or contact lenses. More recently, it is reported that the children wearing orthok lens of smaller back optical zone diameter (BOZD) demonstrated a smaller axial elongation when compared to children wearing lens with larger BOZD. We aimed to explored the myopia efficacy and visual quality of ortho-k with different BOZD (5.0mm or 6.2mm).

DETAILED DESCRIPTION:
This prospective study aimed to evaluate the efficacy of orthokeratology lenses with different back optical zone diameters (BOZD) in slowing axial elongation. Additionally, visual quality will be assessed through measurements of wavefront aberrations, contrast sensitivity, and subjective visual quality using a validated questionnaire. The study seeks to explore the effectiveness of various Ortho-K lens designs and the potential factors influencing their outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age between 8 and 13 years.
* Subjective refraction under cycloplegia: spherical power between -4.00 D and
* 1.00 D, with cylindrical power≤ 1.50 D.
* Best-corrected visual acuity (BCVA) of ≥ 1.0 based on subjective refraction.
* Willing to participate in the clinical trial and provide signed informed consent.

Exclusion Criteria:

* One eye met the inclusion criteria
* Patients with systemic diseases causing immunocompromised or affecting orthokeratology
* There are other eye diseases that affect orthokeratology lens wearing, such as dacryocystitis, blepharitis, various inflammation, glaucoma, etc
* Abnormal cornea
* Previous corneal surgery or corneal trauma history
* Active keratitis (e.g., corneal infection)
* Patients with best corrected distance visual acuity of less than 5.0
* Patients with corneal flat curvature lower than 39.00D, or higher than 48.00D
* Patients with refractive instability
* Patients with overt strabismus
* The corneal epithelium showed obvious fluorescent staining, which was not suitable for patients wearing orthokeratology lenses
* Patients with dry eye are not suitable for orthokeratology
* Patients with corneal endothelial cell density less than 2000 cells /mm2
* Patients who had worn rigid contact lenses (including orthokeratology lenses) within the previous 30 days

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Changes in axial length | The change of baseline and 1years
  Axial length was measured with a biometer

OTHER OUTCOMES:
Change of visual quality | Follow-up evaluations were conducted at baseline, and at 1 day, 1 week, 1 month, 3 months, 6 months, and 12 months after lens wear. The differences from baseline were calculated for each follow-up period.
  The visual quality questionnaire used in this study was adapted from the questionnaire developed by Tilia et al. The questionnaire comprises five categories with a total of nine questions, each accompanied by descriptive text and illustrative images to assist participants in providing their responses. Participants were asked to select the image corresponding to each question, and their responses were converted into numerical scores ranging from 1 to 10, where a score of 1 represents the poorest visual quality.
Change of wavefront aberrations | Follow-up evaluations were conducted at baseline, and at 1 day, 1 week, 1 month, 3 months, 6 months, and 12 months after lens wear. The differences from baseline were calculated for each follow-up period.
  Wavefront aberration data for the eye were obtained using a Hartmann-Shack wavefront sensor (i.Profiler plus, Carl Zeiss Co., Aalen, Germany). The data were analyzed using Zernike polynomial decomposition to calculate the root mean square (RMS) values of total higher-order aberrations (HOAs), spherical aberration, coma aberration, trefoil, astigmatism, and fourth-order aberrations.
Change of contract sensitivity | Follow-up evaluations were conducted at baseline, and at 1 week, 1 month, 3 months, and 12 months after lens wear. The differences from baseline were calculated for each follow-up period.
  Contrast sensitivity was assessed using the OPTEC 6500P contrast sensitivity tester (OPTEC 6500P, Stereo Optical Company, Inc., Chicago, USA) at five spatial frequencies: 1.5, 3, 6, 12, and 18 cycles/degree. The contrast sensitivity scores were expressed in logarithmic units (base 10) following a logarithmic transformation.

CONTACTS AND LOCATIONS:
Overall Officials: Tianjin Eye Hospital, Principal Investigator — Tianjin Eye Hospital Opotometic Center
Locations (1):
- Tianjin Eye Hospital Opotometric Center, Tianjin, Tianjin Municipality, China